CLINICAL TRIAL: NCT03693261
Title: Epicardial Fat as Brown Fat in Coronary Artery Disease
Brief Title: Epicardial Fat in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gianluca Iacobellis, Professor of Medicine, University of Miami
Other Study IDs: 20110879
Record Dates: First submitted 2018-09-30; First posted 2018-10-02 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
Keywords: epicardial fat
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass; Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Adipose tissue will be collected during the cardiac surgery. Epicardial adipose tissue (EAT) biopsy samples (average 0.5-1.0 g) will be taken by cardiac surgeon after anesthesia, before heparin administration, near the proximal tract of the right coronary artery. Each tissue sample will be snap frozen in liquid nitrogen and stored at -80 °C until analysis in a freezer . The subcutaneous fat tissue (SAT) will be harvested at the site of the thoracic wound and preserved in the same manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary Artery Disease (CAD): Patients with clinically and angiographically established coronary artery disease (CAD) who require CABG, as part of the standard medical care.
  Interventions: Procedure: Coronary artery bypass grafting (CABG)
- controls: Control group will be formed by subjects, randomly selected, who will undergo cardiac surgery for aortic or mitral valve replacement as part of their standard medical care (these patients have no history, clinical signs of CAD, and show normal coronary arteries on coronary angiography).
  Interventions: Procedure: Valve replacement

INTERVENTIONS:
Procedure: Coronary artery bypass grafting (CABG) — CABG, as part of the standard medical care
  Groups: Coronary Artery Disease (CAD)
Procedure: Valve replacement — cardiac surgery for aortic or mitral valve replacement as part of their standard medical care
  Groups: controls

SUMMARY:
We hypothesize that human epicardial fat plays a thermogenic role to the myocardium. We hypothesize that epicardial fat may express genes of brown fat and thyroid function that are down-regulated by the presence of coronary artery disease. Because the postulated metabolic role of the epicardial fat, we also hypothesize that the gene expression of these regulatory thermogenic factors is higher in epicardial than subcutaneous fat

This will be a cross-sectional study conducted over a one-year period in patients with or without coronary artery disease who require elective cardiac surgery regardless their participation in the study.

Study group will be formed by 50 patients with clinically and angiographically established CAD who will undergo coronary artery bypass graft, as part of their standard medical care. Control group will be formed by 10 subjects, randomly selected, who will undergo cardiac surgery for aortic or mitral valve replacement as part of their standard medical care (these patients have no history, clinical signs of CAD, and show normal coronary arteries on coronary angiography).

This will be a cross-sectional study conducted over a one-year period in patients with or without coronary artery disease who require elective cardiac surgery regardless their participation in the study.

Adipose tissue will be collected during the cardiac surgery.

DETAILED DESCRIPTION:
Our previous studies indicate that epicardial fat, the visceral fat depot of the heart, plays a role in modulating the heart morphology and its function (Iacobellis et al 2005). Notably, no muscle fascia divides the epicardial fat and the myocardium and the two tissues share the same microcirculation (Iacobellis et al 2005). Epicardial fat has peculiar biochemical properties and is actively involved in lipid and energy homeostasis. Epicardial fat is also a source of several bioactive molecules that might directly influence the myocardium and coronary arteries (Iacobellis et al, 2005,). Because of its anatomic proximity to the myocardium and its intense paracrine and metabolic activity, it is suggested that epicardial fat cytokines reach the myocardium through paracrine or vasocrine pathways and consequently modify its function. Given all these effects and properties, epicardial fat is pathophysiologically and clinically related to development and progression of coronary artery disease and atherosclerosis, regardless of obesity (Iacobellis 2010). Additionally, epicardial fat directly correlates with the intramyocardial lipid content, as we recently described (Malavazos 2010), suggesting a real interaction between the two tissues. However, a dichotomous role has been actually attributed to the epicardial fat. In fact, under physiological conditions epicardial fat displays cardioprotective effects (Iacobellis 2009) and potentially energetic and thermogenic properties, as brown fat (Sacks 2009). Although the interpretation of this finding is still unclear, expression of uncoupling protein1 (UCP1), a marker of brown fat, has been found in human epicardial fat and significantly higher than in subcutaneous fat. We know that brown fat generates heat in response to cold temperatures and activation of the autonomic nervous system under the direct control of thyroid hormones (Bianco 2011). Although the interest in brown fat in humans is growing, our understanding of its actual role in humans is still unclear. The heart is a highly demand organ, under the metabolic control of the thyroid and possibly the epicardial fat. Interestingly experimental models show that hypoxia induces type 3 deiodinase (D3) overexpression in the myocardium that inactivates T3 during ischemia, to protectively decrease cardiomyocytes metabolism and energy expenditure (Simonides et al 2008). Epicardial fat may function like brown fat and thyroid target tissue to protect and defend the myocardium and coronary artery against hypothermia and chronic hypoxia. Nevertheless, whether epicardial fat may have this role and whether this may be affected by the presence of coronary artery disease is currently unknown. We therefore hypothesize that human epicardial fat plays a thermogenic role to the myocardium. We hypothesize that epicardial fat may express genes of brown fat and thyroid function that are downregulated by the presence of coronary artery disease. Because the postulated metabolic role of the epicardial fat, we also hypothesize that the gene expression of these regulatory thermogenic factors is higher in epicardial than subcutaneous fat. These hypotheses will be tested as follows:Specific Aims Ia)Does human epicardial fat express makers of brown adipose tissue, such UCP1 and brown adipocyte differentiation transcription factors in subjects with and without coronary artery disease?b)Does human epicardial fat express type 2 and type 3 deiodinase, thyroid hormones and 3 adrenergic receptors in subjects with and without coronary artery disease?c)Is the thermoregulatory function of the human epicardial fat correlated to the presence and severity of coronary artery disease? Specific Aims IIa)Does the expression of brown fat and thyroid markers gene expression is higher in epicardial than subcutaneous fat?b)Does epicardial fat thickness, as measured by echocardiography, correlate with the gene expression of brown adipose tissue and thyroid markers?c)Does epicardial fat thickness, as measured by echocardiography, correlate with the presence and severity of coronary artery disease?

ELIGIBILITY:
Inclusion Criteria:

Subjects with clinically and angiographically established CAD

Controls: subjects with have no history, clinical signs of CAD, and show normal coronary arteries on coronary angiography, who will undergo cardiac surgery for aortic or mitral valve replacement as part of their standard medical care

Exclusion Criteria:

Patients with heart failure, kidney failure or liver failure, infective disease or cancer will be excluded from the study. Subjects taking glucocorticoids or estrogens or patients currently smoking will be excluded from the study. Patients with mental disorders will also not be included

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The total number of patients participating in the research will be 60. The study group will be formed by 50 consecutive patients, male and female, age 50-75 years, Caucasian, Hispanic and African American, patients with clinically and angiographically established CAD who will undergo CABG, as part of their standard medical care. The control group will be formed by 10 subjects male and female age 50-75 years, randomly selected, who will undergo cardiac surgery for aortic or mitral valve replacement as part of their standard medical care; these patients have no history, clinical signs of CAD, and show normal coronary arteries on coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-12-18 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
EAT thermoregulatory genes | 24 hours
  Does human epicardial fat express makers of brown adipose tissue, such UCP-1 and brown adipocyte differentiation transcription factors in subjects with and without coronary artery disease? Does human epicardial fat express type 2 and type 3 deiodinase, thyroid hormones and β-3 adrenergic receptors in subjects with and without coronary artery disease? Is the thermoregulatory function of the human epicardial fat correlated to the presence and severity of coronary artery disease?

SECONDARY OUTCOMES:
Subcutaneous fat genes | 24 hours
  Does the expression of brown fat and thyroid markers gene expression is higher in epicardial than subcutaneous fat?

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided